CLINICAL TRIAL: NCT01937988
Title: Patient Support During Surgical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2246
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Surgical Abortion
Keywords: Doula; Abortion; Pain; support
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doula Arm (Experimental): Women in the doula arm will have standard procedure protocol with addition of doula support at the time of the procedure.
  Interventions: Other: Doula Arm
- Control Group (No Intervention): Women in the control arm will have standard procedure protocol at the time of the procedure.

INTERVENTIONS:
Other: Doula Arm
  Arms: Doula Arm

SUMMARY:
This study will be a non-blinded randomized controlled trial (RCT) of women presenting for abortion at <13 6/7 weeks. Women will be randomized either to receive support by a trained abortion doula (intervention) or to have standard procedure (control) during the abortion procedure. The investigators hypothesize that women who receive doula support during a first trimester abortion will report less pain during the abortion procedure compared to women who do not receive abortion doula support.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Gestational age by sonogram < 13 6/7 weeks gestation
* Desires pregnancy termination
* Ability to understand the study and give informed consent
* Ability to read and comprehend informed consent document in English

Exclusion Criteria:

* Aged < 18 years
* Gestational age by sonogram > 13 6/7 weeks gestation
* Inability to understand the study and give informed consent
* Inability to read and comprehend informed consent document in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain at time of procedure | At time of procedure
  To determine the effect of abortion doula support during a 1st trimester abortion (< 13 6/7 wks gestational age) on the pain at the time of the abortion, as measured using a 100-mm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Satisfaction with procedure | 10 minutes post-procedure
  To assess the impact of abortion doula support on a woman's overall satisfaction with the abortion experience, as measured using a 100-mm Visual Analog Scale (VAS)
Difficulty of procedure | Immediately post-procedure
  To assess the impact of abortion doula support on the provider's assessment of difficulty of procedure, as measured using a 4-point Likert scale.
Duration of procedure | During procedure
  To assess the impact of doula support on the duration of the procedure, from placement of the speculum to removal of the speculum upon completion of the procedure.
Pain at time of speculum insertion | At time of speculum insertion
  To determine the effect of abortion doula support during a 1st trimester abortion on the pain at the time of speculum insertion, as measured using a 100-mm Visual Analog Scale (VAS).
Anticipated pain | Prior to procedure
  To assess pain anticipated prior to procedure, as measured using a 100-mm Visual Analog Scale (VAS).
Pre-procedure anxiety | Prior to procedure
  To assess anxiety prior to procedure, as measured using a 100-mm Visual Analog Scale (VAS).
Post-procedure recalled pain | Post-procedure
  To assess recalled pain 10 minutes post-procedure, as measured using a 100-mm Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois, United States